CLINICAL TRIAL: NCT03981926
Title: Team-Based Connected Health (TCH) to Improve Clinical Outcomes and Access in Atopic Dermatitis
Acronym: TCH in AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, April Armstrong, Professor and Chief of Dermatology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-16-00914; 1R01AR073486-01A1 (NIH)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis Eczema; Atopic Dermatitis; Eczema
Keywords: Telemedicine; Pragmatic; Equivalency; Skin diseases
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Skin Diseases

STUDY DESIGN:
Intervention Model Description: This is a pragmatic, randomized, controlled, equivalency trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person (No Intervention): In-person care is the control group because it is currently considered the standard of care in delivering dermatologic services. The intervention includes regular visits to a physician, and may include such treatments as ointments, steroids or ultraviolet therapy at the discretion of a physician. In-person care is the major healthcare-delivery model for managing chronic skin diseases and a realistic, primary option that patients face. The patients in the in-person arm can seek atopic dermatitis care from primary care practitioners or dermatologists, just as they would in the real world.
- Team-Based Connected Health (TCH) (Experimental): The intervention arm is the team-based connected health (TCH) model, which purports to increase access to specialists and improve outcomes. Specifically, TCH offers multiple modalities for patients and primary care providers (PCPs) to access dermatologists online directly and asynchronously. TCH also fosters team care and patient engagement through active sharing of management plans and multidirectional, informed communication among patients, PCPs, and dermatologists.
  Interventions: Other: Team-Based Connected Health (TCH)

INTERVENTIONS:
Other: Team-Based Connected Health (TCH) — TCH is an asynchronous, secure online platform where patients can upload images of atopic dermatitis disease and submit assessments. Likewise, practitioners can request and/or initiate dermatology consultations, assume longitudinal care or communicate with patients directly.
  Other Names: Online healthcare; Teledermatology
  Arms: Team-Based Connected Health (TCH)

SUMMARY:
This is a pragmatic, randomized, controlled, equivalency trial. This 12-month trial will evaluate the impact of an online, team-based connected health (TCH) model for management of atopic dermatitis (AD) as compared to in-person care. 300 patients will be randomly assigned to the online TCH model or the in-person control arm. This pragmatic, randomized trial will compare AD disease severity (Aim 1), quality-of-life and access-to-care measures (Aim 2), and costs (Aim 3) between the two models.

DETAILED DESCRIPTION:
Skin diseases account for 30% of all physician office visits. In the United States, access to dermatologists remains a significant challenge for those in underserved or rural communities. To increase access to specialists and improve patient outcomes, we will evaluate a team-based connected health (TCH) model that enables structured asynchronous online interactions among patients, primary care providers (PCPs), and dermatologists. The goal of TCH is to enable effective management of chronic skin diseases via high-quality and efficient online care between providers and patients. TCH purports to bring direct and expedient specialist care to patients and PCPs in a location-independent and asynchronous manner.

Specifically, TCH offers several ways that patients and providers can communicate online asynchronously to manage skin diseases: (1) PCP-dermatologist, (2) patient-dermatologist, and (3) patient-PCP interactions. With PCP-dermatologist interactions, PCPs can access dermatologists online asynchronously for consultations or to request a dermatologist to assume care of the patient's skin disease. With patient-dermatologist interactions, patients can upload clinical images and history online and obtain asynchronous evaluation and recommendations from dermatologists directly. Finally, PCPs have the option of managing their patients' skin diseases online. Importantly, TCH applies efficient workflow that maximally supports providers and fosters multi-directional, informed communication among patients, PCPs, and dermatologists.

To evaluate the impact of TCH, we use atopic dermatitis (AD) as a disease model. AD is a common, relapsing inflammatory skin disease affecting 32 million individuals in the U.S. AD is characterized by intense itching and red, scaly patches. It incurs significant morbidities and high healthcare costs. To address skin inflammation, itch, and psychosocial consequences, PCPs and dermatologists need to adopt a team-based approach to effectively manage all aspects of AD.

The primary goal of the proposed research is to test whether the online TCH model results in equivalent improvements in disease severity and quality of life, provides better access to specialist care, and is cost-saving as compared to usual in-person care in pediatric and adult patients with AD. Specifically, we will conduct a pragmatic, cluster-randomized controlled equivalency trial and use validated measures to compare AD disease severity, health-related quality of life, and access to care between TCH and in-person care. We will also compare costs of the two healthcare delivery models from a societal perspective by conducting cost- minimization and sensitivity analyses.

This proposal evaluates a significant innovation in specialty-care delivery that will likely result in improved patient outcomes, greater access to specialists, and cost savings. The study findings will be highly impactful and have immense dissemination potential to the management of many other chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 year or older
* Physician-diagnosed atopic dermatitis (AD)
* Access to a digital-photo capturing device (mobile phone or camera) capable of capturing images with a minimum resolution of 1024x768 pixels
* Access to internet
* Able to establish care or have established care with providers
* Provision of signed and dated informed consent and youth assent form

Exclusion Criteria:

* Unable to fulfill study-related tasks by adult AD patients or parents or guardians of pediatric AD patients

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: April W Armstrong, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | In-Person | Team-Based Connected Health (TCH)
Started | 151 | 149
Completed | 146 | 140
Not Completed | 5 | 9
Not completed — Lost to Follow-up | 5 | 9

BASELINE CHARACTERISTICS:
Population: A total of 300 patients were enrolled, and 151 patients were randomized to the in-person group and 149 patients were randomized to the online group. Each participant was followed for 12 months. The analyses were based on intention-to-treat.
Groups:
- Total: Total of all reporting groups
Arm/Group | In-Person | Team-Based Connected Health (TCH) | Total
Number analyzed (Participants) | 151 | 149 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (16.6) | 37.2 (18.2) | 34.6 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 105 | 211
  Male | 45 | 44 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 47 | 86
  Not Hispanic or Latino | 110 | 102 | 212
  Unknown or Not Reported | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1 | 0 | 1
  Asian | 65 | 47 | 112
  Black or African American | 12 | 15 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 53 | 63 | 116
  Other | 20 | 23 | 43
Education [Count of Participants; unit: Participants]
  Grades 1-8 (Grade School) | 10 | 11 | 21
  Some High School | 5 | 5 | 10
  High School Diploma or Equivalent (GED) | 7 | 8 | 15
  Some College, No Degree | 26 | 33 | 59
  College Degree | 49 | 54 | 103
  Graduate or Doctoral Degree | 35 | 32 | 67
  Not Applicable | 18 | 6 | 24
  Unknown or Not Reported | 1 | 0 | 1
Insurance Type [Count of Participants; unit: Participants]
  Private or Health Maintenance Organization (HMO) | 111 | 99 | 210
  Medicaid | 20 | 22 | 42
  Medicare | 12 | 20 | 32
  No Insurance | 5 | 7 | 12
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Disease Severity as Measured by the Eczema Area and Severity Index (EASI)
Description: EASI combines the assessment of disease severity (erythema, induration, excoriation, and lichenification) and the affected area into a single score between 0 (no disease) to 72 (maximal disease). The primary outcome of the study is the mean improvement in EASI.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | In-Person | Team-Based Connected Health (TCH)
Number analyzed (Participants) | 151 | 149
score on a scale
  Baseline | 4.81 [4.04 to 5.59] | 4.93 [3.90 to 5.95]
  Month 12 | 2.70 [1.97 to 3.43] | 2.76 [2.16 to 3.35]

2. Secondary Outcome: Change in Disease Severity as Measured by the Validated Investigator Global Assessment (vIGA)
Description: vIGA is an ordinal scale that provides a global assessment of the patient's AD disease severity. vIGA is scored on a 5-point ordinal scale ranging from 0 (clear) to 4 (severe). The overall change in disease severity for this outcome is measured by calculating the change in vIGA score from baseline averaged across 12 months.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | In-Person | Team-Based Connected Health (TCH)
Number analyzed (Participants) | 151 | 149
score on a scale
  Baseline | 2.28 [2.12 to 2.45] | 2.48 [2.30 to 2.65]
  Month 12 | 1.71 [1.55 to 1.86] | 1.56 [1.39 to 1.73]

3. Secondary Outcome: Change in Disease Severity as Measured by the Patient-Oriented Eczema Measure (POEM).
Description: POEM is a 7-item tool for patient and/or proxy self-completion used to monitor atopic dermatitis severity, focusing on the illness as experienced by the patient. Scores range from 0 (clear) to 28 (very severe). The overall change in disease severity for this outcome will be measured by calculating the change in POEM score from baseline averaged across 12 months.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | In-Person | Team-Based Connected Health (TCH)
Number analyzed (Participants) | 151 | 149
score on a scale
  Baseline | 11.7 [10.5 to 12.9] | 11.6 [10.5 to 12.8]
  Month 12 | 8.57 [7.55 to 9.59] | 7.70 [6.65 to 8.74]

4. Secondary Outcome: Change in Quality of Life as Measured by the Dermatology Life Quality Index (DLQI) and the Children's Dermatology Quality Index (CDLQI)
Description: The DLQI and the CDLQI are validated, 10-question questionnaires that can be used to assess dermatology-specific quality of life in adults and children with atopic dermatitis. Scores range from 0 to 30, with higher scores indicating more severe impact on quality of life. The overall change in quality of life for this outcome is measured by calculating the change in DLQI / CDLQI from baseline averaged across 12 months.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | In-Person | Team-Based Connected Health (TCH)
Number analyzed (Participants) | 151 | 149
score on a scale
  Baseline | 7.73 [6.73 to 8.73] | 8.04 [7.00 to 9.08]
  Month 12 | 6.52 [5.46 to 7.58] | 6.10 [5.03 to 7.17]

5. Secondary Outcome: Change in Quality of Life as Measured by the EQ-5D-5L and the EQ-5D-Y
Description: EQ-5D-5L and EQ-5D-Y are validated measures of health status. The EQ-5D-5L and the EQ-5D-Y provide an index value that can be used for quality of life and economic evaluations. An index value of 0 represents a health state equivalent to death and an index value of 1 represents full health. The EQ-5D-5L and the EQ-5D-Y also provide a Visual Analogue Score (VAS) where respondents rate their perceived health from 0 (worst imaginable health) to 100 (best imaginable health). The overall change in quality of life for this outcome is measured by calculating the change in utility index and VAS from baseline averaged across 12 months.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | In-Person | Team-Based Connected Health (TCH)
Number analyzed (Participants) | 151 | 149
score on a scale
  Utility Index Baseline | 0.86 [0.83 to 0.89] | 0.85 [0.82 to 0.88]
  Utility Index Month 12 | 0.87 [0.84 to 0.91] | 0.87 [0.84 to 0.90]
  VAS Baseline | 82.6 [80.2 to 84.9] | 82.0 [80.0 to 84.1]
  VAS Month 12 | 84.2 [82.3 to 86.2] | 84.4 [82.3 to 86.4]

6. Secondary Outcome: Access to Care: Transportation
Description: Access-to-care measures include mode of transportation.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | In-Person | Team-Based Connected Health (TCH)
Number analyzed (Participants) | 151 | 149
Participants
  Bus or Train | 12 | 9
  Car | 131 | 139
  Walking | 7 | 1
  Unknown or Not Reported | 1 | 0

7. Secondary Outcome: Access to Care: Wait Time
Description: Access-to-care measures include time needed for evaluation.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | In-Person | Team-Based Connected Health (TCH)
Number analyzed (Participants) | 151 | 149
minutes
  Baseline | 65.9 (46.1) | 51.6 (39.4)
  Month 12 | 30.1 (33.1) | 29.1 (30.0)

8. Secondary Outcome: Change in Healthcare Utilization and Healthcare Costs: Healthcare Utilization
Description: We will compare differences in healthcare utilization by using the Cornell Services Index (CSI). The CSI is a validated method to assess health service use. Mean time per medical, psychological, and professional visits will be calculated.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | In-Person | Team-Based Connected Health (TCH)
Number analyzed (Participants) | 151 | 149
minutes
  Time per Medical Visit | 44.6 (45.2) | 46.0 (38.1)
  Time per Psychological Visit | 51.1 (13.3) | 45.5 (14.5)
  Time per Professional Visit | 38.1 (22.4) | 36.7 (20.8)

9. Secondary Outcome: Change in Healthcare Utilization and Healthcare Costs: Healthcare Costs
Description: We will compare differences in healthcare costs by using the Cornell Services Index (CSI). The CSI is a validated method to assess health service use. Mean out-of-pocket costs across medical, psychological, and professional visits will be calculated.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | In-Person | Team-Based Connected Health (TCH)
Number analyzed (Participants) | 151 | 149
dollars | 201.7 (701) | 48.3 (45)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | In-Person | Team-Based Connected Health (TCH)
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/149
Serious Adverse Events (participants affected / at risk) | 2/151 | 1/149
Other Adverse Events (participants affected / at risk) | 0/151 | 0/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | In-Person (N=151) | Team-Based Connected Health (TCH) (N=149)
Biliary acute pancreatitis (Gastrointestinal disorders) | 1 | 0
Anaphylaxis (Immune system disorders) | 0 | 1
Tibia fracture (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT03981926/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT03981926/ICF_001.pdf